CLINICAL TRIAL: NCT03319355
Title: The Effect of a 12-week Multicomponent Therapy in Fibromyalgia
Brief Title: Multicomponent Therapy for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: AZ Alma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: EC/EH/111221
Record Dates: First submitted 2017-10-05; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Fibromyalgia
Keywords: multicomponent therapy
MeSH Terms: conditions — Fibromyalgia | interventions — Cognitive Behavioral Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — exercise therapy
  Other Names: physical therapy

SUMMARY:
Therapy for fibromyalgia is a well discussed topic in literature, yet not thoroughly evidence-based. Several unicomponent therapies seem to be benificial. Whereas multicomponent and multidisciplinary therapy gains importance and revealing promising results, the investigators aim to combine two well-known therapies in a program for patients with fibromyalgia.

From clinical experience, a high drop-out rate has been stated. All data will be explored to analyse explanatory factors.

ELIGIBILITY:
Inclusion Criteria:

* woman with fibromyalgia
* between the age of 20 and 50
* agreement with therapy protocol

Exclusion Criteria:

* high indication of depression measured with the Beck Depression Index

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | 6weeks
  impact of fibromyalgia on daily life with a questionnaire
Tampa scale for kinesiophobia | 6weeks
  rating the kinesiophobia with a questionnaire
Beck Depression Index | 6 weeks
  degree of depression with a questionnaire
Pain Coping Inventory | 6 weeks
  inventory of the use of pain coping strategies with a questionnaiire
Pain at tenderpoints | 6 weeks
  measuring tolerable pain at specified tenderpoints with an algometer
Grip strength | 6 weeks
  measuring grip strength of both hands with a dynamometer
Walking | 6 weeks
  6 minute walking test on a treadmill
cycling | 6 weeks
  10 minutes cycling test on a hometrainer

IPD SHARING:
Plan to Share IPD: No